CLINICAL TRIAL: NCT05215236
Title: Prospective, Randomized, Controlled Trial of an Opiate Sparing Protocol Versus Standard Opiate Based Protocol Following Open Reduction Internal Fixation of Distal Radius Fractures
Brief Title: Opiate Sparing Protocol Randomized Controlled Trial in Open Distal Radius Fracture Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, William Jacob Weller, Principal Investigator, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-08332-FB
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opiate Sparing (Experimental): Standard icing and elevation therapy Acetaminophen 1000 milligrams by mouth every 8 hours for five days then as needed every 8 hours for pain control Gabapentin 100 milligrams by mouth three times per day for 14 days Celecoxib 100 milligrams by mouth two times per day for 5 days Esomeprazole 20 milligrams by mouth once per day for 14 days Promethazine 12.5 milligrams by mouth every 8 hours as needed for nausea or vomiting Docusate 100 milligrams by mouth two times per day while taking oxycodone Oxycodone 5 milligrams by mouth every 6 hours as needed for pain control unresponsive to other medications
  Interventions: Other: Opiate Sparing
- Opiate Based (Active Comparator): Standard icing and elevation therapy Oxycodone 5-10 milligrams by mouth every 4 to 6 hours as needed for pain control Acetaminophen 1000 milligrams by mouth every 8 hours as needed for pain control Promethazine 12.5 milligrams by mouth every 8 hours as needed for nausea or vomiting Docusate 100 milligrams by mouth two times per day while taking oxycodone
  Interventions: Other: Opiate Based

INTERVENTIONS:
Other: Opiate Sparing — Subjects will receive non-opiate medications for pain control
  Arms: Opiate Sparing
Other: Opiate Based — Subjects will receive opiate based medications for pain control
  Arms: Opiate Based

SUMMARY:
A comparison of oral morphine equivalents between an opiate sparing cohort and an opiate based cohort following open reduction internal fixation of a distal radius fracture.

DETAILED DESCRIPTION:
Recently, the opioid epidemic has been the center of focus for healthcare providers and governmental agencies due to rising rates of opioid abuse, opioid-related fatalities, and overall economic burden of treating the opioid epidemic. The prescribing patterns of opioid pain medications have fallen under scrutiny and healthcare providers have sought alternative pain management strategies that have limited opioid pain medication use. As orthopaedic surgeons account for 7.7% of all dispensed opioid prescriptions within the United States, surgeons have investigated multimodal pain management strategies to assess effectiveness in controlling postoperative pain as well as limiting opioid use and opioid related complications. The literature documents the safety and effectiveness of non-steroid anti-inflammatory drugs (NSAID) and acetaminophen in soft tissue hand procedures and distal radius fracture plating. Currently, there remains no clear consensus on the ideal pain management strategy following open reduction internal fixation (ORIF) of distal radius fractures and the vast majority of strategies are based on opiate-driven protocols. This study will investigate the effectiveness of an opiate sparing protocol following open reduction and internal fixation (ORIF) of distal radius fractures on opiate consumption as measured by oral morphine equivalents at the 2, 6 and 12 week postoperative time point through collection of pill counts. Secondary outcomes are pain scores, patient satisfaction, and safety reporting (complications, reoperations, and readmissions) during the 12-week episode-of-care. This study will document the safety and effectiveness of an opiate sparing, multimodal pain management protocol in properly selected patients undergoing ORIF of distal radius fractures.

Following written consent documentation, Subjects will be randomized to either the opiate sparing cohort or the opiate based cohort at a 1:1 randomization. No blinding will occur as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Open reduction internal fixation surgery at Campbell Clinic Surgery Center
* Body Mass Index less than or equal to 45
* Fluent in verbal and written English

Exclusion Criteria:

* Known sensitivity to medications in either protocol
* Renal disease by medical history
* Concomitant ipsilateral upper extremity injury or condition other than wrist
* Chronic pain syndrome
* Consumption of ten consecutive day so opioid use in the previous 90 days
* Worker's compensation
* Women who are pregnant, planning to become pregnant, or are breastfeeding
* Takes either angiotensin-converting enzyme inhibitor or angiotensin II receptor blockers for hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Oral Morphine Equivalent | postoperative day to two week visit
  opiate pill count
Oral Morphine Equivalent | two week to six week visit
  opiate pill count
Oral Morphine Equivalent | six week to twelve week visit
  opiate pill count

SECONDARY OUTCOMES:
Visual Analog Score | postoperative day to two week visit
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain
Visual Analog Score | six week visit
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain
Visual Analog Score | twelve week visit
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain

OTHER OUTCOMES:
Incidence of treatment-emergent adverse event | postoperative day to two week visit
  monitoring for safety events
Incidence of treatment-emergent adverse event | two week to six week visit
  monitoring for safety events
Incidence of treatment-emergent adverse event | six week to twelve week visit
  monitoring for safety events
Patient satisfaction Score | postoperative day to two week visit
  patient reported satisfaction with pain management from 0 to 10 where 0 is very unsatisfied and 10 is very satisfied
Patient satisfaction Score | two week to six week visit
  patient reported satisfaction with pain management from 0 to 10 where 0 is very unsatisfied and 10 is very satisfied
Patient satisfaction Score | six week to twelve week visit
  patient reported satisfaction with pain management from 0 to 10 where 0 is very unsatisfied and 10 is very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: William J Weller, MD, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galos DK, Taormina DP, Crespo A, Ding DY, Sapienza A, Jain S, Tejwani NC. Does Brachial Plexus Blockade Result in Improved Pain Scores After Distal Radius Fracture Fixation? A Randomized Trial. Clin Orthop Relat Res. 2016 May;474(5):1247-54. doi: 10.1007/s11999-016-4735-1. Epub 2016 Feb 11. PMID 26869374
- [Background] Martinez L, Ekman E, Nakhla N. Perioperative Opioid-sparing Strategies: Utility of Conventional NSAIDs in Adults. Clin Ther. 2019 Dec;41(12):2612-2628. doi: 10.1016/j.clinthera.2019.10.002. Epub 2019 Nov 14. PMID 31733939
- [Background] Niedermeier SR, Crouser N, Hidden K, Jain SA. Pain Management following Open Reduction and Internal Fixation of Distal Radius Fractures. J Wrist Surg. 2021 Feb;10(1):27-30. doi: 10.1055/s-0040-1716508. Epub 2020 Oct 14. PMID 33552691
- [Background] O'Neil JT, Wang ML, Kim N, Maltenfort M, Ilyas AM. Prospective Evaluation of Opioid Consumption After Distal Radius Fracture Repair Surgery. Am J Orthop (Belle Mead NJ). 2017 Jan/Feb;46(1):E35-E40. PMID 28235120
- [Background] Padilla JA, Gabor JA, Schwarzkopf R, Davidovitch RI. A Novel Opioid-Sparing Pain Management Protocol Following Total Hip Arthroplasty: Effects on Opioid Consumption, Pain Severity, and Patient-Reported Outcomes. J Arthroplasty. 2019 Nov;34(11):2669-2675. doi: 10.1016/j.arth.2019.06.038. Epub 2019 Jun 26. PMID 31311667
- [Background] Sabatino MJ, Kunkel ST, Ramkumar DB, Keeney BJ, Jevsevar DS. Excess Opioid Medication and Variation in Prescribing Patterns Following Common Orthopaedic Procedures. J Bone Joint Surg Am. 2018 Feb 7;100(3):180-188. doi: 10.2106/JBJS.17.00672. PMID 29406338
- [Background] Thybo KH, Hagi-Pedersen D, Dahl JB, Wetterslev J, Nersesjan M, Jakobsen JC, Pedersen NA, Overgaard S, Schroder HM, Schmidt H, Bjorck JG, Skovmand K, Frederiksen R, Buus-Nielsen M, Sorensen CV, Kruuse LS, Lindholm P, Mathiesen O. Effect of Combination of Paracetamol (Acetaminophen) and Ibuprofen vs Either Alone on Patient-Controlled Morphine Consumption in the First 24 Hours After Total Hip Arthroplasty: The PANSAID Randomized Clinical Trial. JAMA. 2019 Feb 12;321(6):562-571. doi: 10.1001/jama.2018.22039. PMID 30747964